CLINICAL TRIAL: NCT07257601
Title: The Effect of Transcranial Direct Current Stimulation Combined With Repetitive Transcranial Magnetic Stimulation on Motor Function Rehabilitation in Patients With Locked-in Syndrome
Brief Title: TDCS-RTMS Intervention for Motor Function
Acronym: TRIMLiS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Qiuyou Xie, principal investigator, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L20251115
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Locked in Syndrome
MeSH Terms: conditions — Locked-In Syndrome | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): true tDCS and true rTMS
  Interventions: Device: Repetitive transcranial magnetic stimulation; Device: Transcranial direct current stimulation
- Group 2 (Placebo Comparator): sham tDCS and true rTMS
  Interventions: Device: Repetitive transcranial magnetic stimulation; Device: Transcranial direct current stimulation
- Group 3 (Placebo Comparator): true tDCS and sham rTMS
  Interventions: Device: Repetitive transcranial magnetic stimulation; Device: Transcranial direct current stimulation
- Group 4 (Placebo Comparator): sham tDCS and sham rTMS
  Interventions: Device: Repetitive transcranial magnetic stimulation; Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — The stimulation intensity is determined by the individual resting motor threshold (RMT), which is the lowest TMS intensity that the target muscle (such as abductor pollicis brevis) can produce EMG signals with peak to peak values greater than 50 μ V at least 5 times in 10 stimuli by stimulating the motor cortex (M1 area). The actual stimulus intensity was 90% of RMT. Using an 8-shaped coil, locate the M1 area on both sides successively (left side in the morning and right side in the afternoon, in the same order as tDCS). Each treatment included 1600 pulses, 4 seconds of stimulation, with an interval of 26 seconds. Each hemisphere was stimulated once a day for 5 consecutive working days. The unilateral M1 area was stimulated 20 times for 4 weeks, and each stimulation lasted 20 minutes. The real rTMS group and the sham rTMS group were treated with the same regimen. The coil was placed 90 degrees perpendicular to the scalp surface with the same parameters as the active rTMS.
  Other Names: rTMS
Device: Transcranial direct current stimulation — Deliver 2mA DC power through a 5 × 5 cm ² sponge electrode, with the anode placed in the M1 area on one side (left side in the morning and right side in the afternoon) and the cathode placed on the opposite shoulder. Each tDCS treatment lasts for a fixed time of 20 minutes throughout the day, approximately 20 minutes before rTMS treatment, five days a week, with a total of 20 sessions in the unilateral M1 area for a total of 4 weeks. The true tDCS group and the false tDCS group received the same treatment plan. For the false tDCS group, patients felt electrical stimulation within 30 seconds, and then the current gradually decreased to 0mA.
  Other Names: tDCS

SUMMARY:
This study was a multicenter randomized double-blind, sham controlled trial initiated by Zhujiang Hospital of Southern Medical University. It is planned to recruit 72 eligible patients with atresia syndrome and randomly divide them into four groups according to the ratio of 1:1:1:1. Group 1 received the sequential stimulation of true tDCS and true rTMS, group 2 received the stimulation of sham tDCS and then true rTMS, group 3 received the stimulation of true tDCS and then sham rTMS, and group 4 received the simulated stimulation of sham tDCS and sham rTMS. The patients were treated for 4 weeks, 5 days a week, once a day in the bilateral M1 area, and in the morning and afternoon on the left and right sides respectively. Each tDCS and rTMS treatment lasted for 20 minutes.Various indicators were evaluated before and after the intervention, and the observation and follow-up were conducted 1, 3, and 6 months after the intervention.

DETAILED DESCRIPTION:
This study was a multicenter randomized double-blind, sham controlled trial initiated by Zhujiang Hospital of Southern Medical University. It is planned to recruit 72 eligible patients with atresia syndrome and randomly divide them into four groups according to the ratio of 1:1:1:1. Group 1 received the sequential stimulation of true tDCS and true rTMS, group 2 received the stimulation of sham tDCS and then true rTMS, group 3 received the stimulation of true tDCS and then sham rTMS, and group 4 received the simulated stimulation of sham tDCS and sham rTMS. The patients were treated for 4 weeks, 5 days a week, once a day in the bilateral M1 area, and in the morning and afternoon on the left and right sides respectively. Transcranial direct current stimulation (tDCS) was performed using a 2 Ma DC stimulator. The anode was placed in the M1 area of the target side (corresponding to the electrode position c3/c4 of the 10-20 EEG system), and the cathode was placed on the contralateral shoulder. The left side was done in the morning and the right side was done in the afternoon. Each tDCS treatment lasted for 20 minutes. The sham stimulation was given current stimulation for 30 seconds and gradually decreased to 0. Repetitive transcranial magnetic stimulation (rTMS) intervention was performed 20 minutes after the end of TDCS treatment. RTMS uses an 8-shaped coil placed in the M1 area of the target side to stimulate at a frequency of 10Hz. Each treatment contains 1600 pulses of stimulation for 4 seconds, with an interval of 26 seconds. The total number of pulses is 1600, lasting for 20 minutes. Each time is once a day in the M1 area of both sides. The sequence is the same as that of TDCS, 5 days a week, and the same lasts for 4 weeks. The stimulation coil was placed at 90 degrees during sham stimulation. Various indicators were evaluated before and after the intervention, and the observation and follow-up were conducted 1, 3, and 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The patients were 18-70 years old, clinically diagnosed as classic or incomplete atresia syndrome, and the onset time was 6 weeks-1 year.
* Clear consciousness, effective communication and command response through eye movement or other established methods.
* No drugs (sodium, calcium channel blockers or sedatives) that may affect neuromuscular function or brain stimulation effect were used, or the drugs were stably stopped for more than 1 week before enrollment.
* The patient or his legal guardian signed the informed consent form and agreed to cooperate in completing all test procedures and evaluations.

Exclusion Criteria:

* Metal implants (such as cardiac pacemaker, intracranial metal clip, etc.), electronic equipment or other TMS contraindications.
* Complicated with severe cognitive impairment (such as dementia) or unable to cooperate to complete the assessment scale test.
* Have a history of severe cardiopulmonary dysfunction, mental illness and seizures.
* There are other neurodegenerative diseases that affect the recovery of motor function (such as amyotrophic lateral sclerosis, etc.)
* Recently (within 1 month) participated in other clinical trials related to neuromodulation therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
the efficiency | Before intervention, 1-2 days after intervention, and 1, 3, and 6 months after intervention
  An increase of 5 points in the Fugl Meyer Assessment (FMA) score or an increase of one level in the House Brackmann Facial Nerve Grading Scale (HBFNGS) score is considered effective through behavioral assessment.

SECONDARY OUTCOMES:
FMA | Before intervention, 1-2 days after intervention, and 1, 3, and 6 months after intervention
  FMA comprehensively covers the assessment of upper and lower limb motor function. In the upper limbs, a detailed assessment was conducted on the motor abilities of the shoulders, elbows, wrists, and hands, including joint range of motion, muscle strength, coordination, and fine motor control.
HBFNGS | Before the intervention starts, 1-2 days after the intervention ends, and 1, 3, and 6 months after the intervention ends
  It is a specialized assessment scale for facial nerve injury, which divides facial nerve function into six levels, from normal to complete paralysis, and provides a detailed grading evaluation of the motor function of facial expression muscles. It has important application value in the diagnosis, treatment effect evaluation, and prognosis judgment of facial nerve injury.
Modified Barthel Index | Before intervention, 1-2 days after intervention, and 1, 3, and 6 months after intervention
  Contains 10 activities of daily living (ADLs), including eating, dressing, toileting, personal hygiene, bathing, bed and chair transfer, walking/wheelchair use, going up and down stairs, bowel control, and urination control. The score for each activity is determined by the level of assistance required by the patient to complete the activity, with a maximum score of 10 points. The total score range is 0-100 points.
Motor evoked potential（Mep） | Before intervention, 1-2 days after intervention
  By transcranial magnetic stimulation or electrical stimulation of the cerebral motor cortex, the excitation of cortical motor neurons is triggered, and the generated electrical impulses are transmitted along the corticospinal tract to the anterior horn motor neurons of the spinal cord, thereby causing corresponding muscle contractions and recording potential changes on the muscle surface. In practical operation, the stimulation electrode is usually placed in a specific motor cortex area of the scalp, while the recording electrode is placed in the muscle belly of the target muscle.
Assessment of TMS-EEG（TEPs） | Before intervention and 1-2 days after intervention
  TEPs refer to the potential changes generated by the synchronous discharge of cortical neurons after TMS pulse stimulation. These potential changes can be recorded through EEG and synchronized with the timing of TMS pulses. TEPs can be used to study the brain's response to stimuli, such as studying the brain's response to different types of TMS stimuli, as well as studying the brain's response to different stimulus intensities. The morphology and amplitude of TEPs can provide information about the activation and inhibition of cortical neurons in the brain.
Assessment of TMS-EEG（oscillation analysis） | Before intervention and 1-2 days after intervention
  Oscillations refer to the oscillations generated by synchronous firing of cortical neurons after TMS pulse stimulation. These oscillations can be recorded by EEG and synchronized with the time of TMS pulses. TMS triggered oscillations can be used to study the brain's response to stimuli of different frequencies, such as studying the brain's response to TMS stimuli of different frequencies, as well as studying the brain's response to sound or light stimuli of different frequencies. The frequency and amplitude of TMS triggered oscillations can provide information about the activation and inhibition of cortical neurons in the brain, as well as the brain's response to different types of stimuli.